CLINICAL TRIAL: NCT01212354
Title: Phase III A Prospective, Randomized, Rater-blinded, Multicentre Interventional Clinical Trial. Do Selective Radiation Dose Escalation and Tumour Hypoxia Status Impact the Locoregional Tumour Control After Radiochemotherapy of Head & Neck Tumours?
Brief Title: Impact of Selective Radiation Dose Escalation and Tumour Hypoxia Status on Locoregional Tumour Control After Radiochemotherapy of HNT
Acronym: Escalox
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESC-928-MOL-0000-I
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Locally Advanced Head and Neck Cancer
Keywords: intensity modulated radiotherapy; selective dose escalation; hypoxia; head cancer; neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Hypoxia | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - experimental (Experimental): 7 weeks Radiotherapy Intervention with with 5x2.3 Gy per week up to a total dose of 80.5 Gy and parallel chemotherapy of 20 mg/m²/d Cisplatin in week 1 and 5.
  Interventions: Radiation: Radiotherapy
- B - control (Active Comparator): 7 weeks Radiotherapy Intervention with 5x2.0 Gy per week up to a total dose of 70 Gy and parallel chemotherapy of 20 mg/m²/d Cisplatin in week 1 and 5.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — 7 weeks Radiation dose escalation (5 x 2.3 Gy up to 80.5 Gy total dose)
  Other Names: IMRT-SIB

SUMMARY:
The major clinical problem and predominant cause of death after radio-oncological treatment of H+N cancers are loco-regional relapses. This randomized trial tests the hypothesis that dose escalated Intensity Modulated Radiotherapy (IMRT) selectively applied to the macroscopic primary tumor and involved neck nodes - which both in 80% - are hypoxic improves loco-regional control by at least 15% at 2 years. IMRT is combined with concurrent Cis-Platin chemotherapy. Tumor volume which correlates with number of malignant cells as well as tumor hypoxia are important biological parameters which increase radio-resistance, failure of local control and tumor progression. Basing on data of experimental and clinical radiation oncology we consider hypoxia as a useful parameter for pre-therapeutic strati-fication in future randomized radio-chemotherapy trials.

In addition, hypoxia imaging by PET can be used for testing the significance of selective dose escalation on hypoxic tumor sub-volumes ("Dose Painting").

As a prerequisite for such innovative studies addressing hypoxia the translational part investigates the following key issues: correlation between the size of total tumor volume (primary, lymph nodes) and hypoxic sub-volume, the spatial shift of the hypoxic sub-volume before start of treatment and the correlation of loco-regional control and hypoxia.

Before starting the main study a pre-study to assess the occurrence of radiation induced toxicities is mandatory to be performed. In a step-wise dose-escalation in a cohort-design the safety of dose-escalation should be determined. Step one: 6 patients Step two: 14 patients. In the pre-study the 1st group (6 patients) should be treated with 2.2 Gy up to 77.0 Gy for DEVPT and DEVLK. After evaluation of the toxicity the next 14 patients should be treated by this scheme.

DETAILED DESCRIPTION:
The pre-study with sequential design is a prospective multicentre interventional pilot study to assess toxicity of intensity modulated radiotherapy (IMRT) plus Cisplatin of head and neck cancers

The main study is a multicenter phase III randomized trial on the effect of dose escalated radiotherapy with concomitant chemotherapy to treat local advanced head and neck cancer. The study compares two treatment arms:

Experimental intervention (group A): 7 weeks standard radio-chemotherapy with 20 mg/m²/d Cisplatin in week 1 and 5 including simultaneous radiation dose escalation (5x2.3 Gy per week up to 80.5 Gy total dose) to the primary tumour and involved neck nodes ≥ 2 cm.

The Dose Escalated tumour Volume (DEVPT) is defined by the macroscopic (Gross) primary Tumour Volume (GTVPT) minus a 3 mm margin at organs at risk or at mucosal sites to reduce the risk of high dose deposition at the surrounding normal tissue. All involved lymph nodes visualized by CT with a minimal diameter of 2 cm are also included for dose escalation (DEVLN). The DEVLN of the lymph nodes > 2 cm is determined by the involved lymph node volume (GTVLN) minus a margin of 3 mm at organs at risk or mucosal sites. The 3 mm margin as well as the part of the target volume with suspected microscopic tumor extension receives 2 Gy per fraction.

Control intervention (group B): 7 weeks standard radio-chemotherapy with 5x2.0 Gy per week up to a total dose of 70 Gy and 20 mg/m²/d Cisplatin in week 1 and 5.

In group A and B: The treatment of the elective cervical lymphatic areas is given in the same session as the GTV but with a single dose of 1.6 Gy up to 56 Gy (so called simultaneous integrated boost concept).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age ≥ 18 ≤ 70 years
* Independent of gender
* Independent of race
* ECOG 0 - 2
* Tumor of oral cavity, oropharynx or hypopharynx
* Histology: squamous cell carcinoma
* Curative treatment intended
* Tumor is classified as irresectable (see Appendix)
* Woman of child-bearing age: negative pregnancy test in serum
* Contraception in male and female patients and their partners if of childbearing potential, willingness to use effective contraceptive method for the study duration and 2 months post therapy
* Sufficient bone marrow reserves during 7 days before study inclusion; (leukocytes ≥ 4 x 109/l, absolute no. of neutrophiles (ANC) ≥ 2 x 109/; thrombocyte count ≥ 100 x 109/l; Hemoglobin ≥ 10g/dl)
* adequate liver function during 7 days before study inclusion (total bilirubine ≤ 2,5 x ULN (upper limit of normal), ASAT/ ALAT ≤ 2,5 x ULN, alkaline phosphatase ≤ 2,5 x ULN of the institution's normal value)
* adequate kidney function during 7 days before study inclusion; serum creatinine ≤ 130 μmol/l; creatinine clearance ≥ 70 ml/min
* all patients should have a dental examination before starting therapy and when necessary be treated, adaptation of a teeth protection bar
* a percutane feeding tube should be applied before start of treatment

Exclusion Criteria:

* Infiltration of the mandible and / or larynx
* impaired renal and/ or liver function
* secondary malignancy, unknown primary cancer, nasopharynx cancer or salivary gland cancers
* Metastatic disease
* Another cancer within 5 years of study entry
* Serious concomitant disease or medical condition
* Pregnancy or lactation
* Women of child-bearing potential with unclear contraception (post menopausal women must have been amenorrheal for at least 12 months to be considered of non-childbearing potential)
* previous treatment with chemotherapy, radiotherapy or surgery in head and neck (except an excisional biopsy or biopsy for histology)
* concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to study screening
* life expectancy of < 12 months
* contraindications to receive Cisplatin
* social situations that limit compliance with study requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2015-07; Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
2 year-loco-regional control | 2 years

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
Progression-free survival (PFS) | 2 years
Time to progression (TTP) | 5 years
Distant metastases (DM) | 2 years
Acute and late toxicity esp. concerning salivary glands | 5 years
Quality of life (EORTC QoL-C30, H&N 35) | 2 years
Adverse effects according to NCI CTC-AE (VERSION 4.0/ 10/1/2010) and LENT-SOMA | 2 years
FMISO PET/CT: Reproducibility and correlation with treatment coutcome | 2 years
Relapse free Survival (RFS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steffi U. Pigorsch, Dr. med., Principal Investigator — Klinik für Strahlentherapie und Radiologische Onkologie, Klinikum rechts der Isar der TU München Ismaningerstr. 22; 81675 Munich, Germany
Locations (1):
- Klinik für RadioOnkologie Strahlentherapie, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Pigorsch SU, Kampfer S, Oechsner M, Mayinger MC, Mozes P, Devecka M, Kessel KK, Combs SE, Wilkens JJ. Report on planning comparison of VMAT, IMRT and helical tomotherapy for the ESCALOX-trial pre-study. Radiat Oncol. 2020 Nov 2;15(1):253. doi: 10.1186/s13014-020-01693-2. PMID 33138837
- [Derived] Pigorsch SU, Wilkens JJ, Kampfer S, Kehl V, Hapfelmeier A, Schlager C, Bier H, Schwaiger M, Combs SE. Do selective radiation dose escalation and tumour hypoxia status impact the loco-regional tumour control after radio-chemotherapy of head & neck tumours? The ESCALOX protocol. Radiat Oncol. 2017 Mar 1;12(1):45. doi: 10.1186/s13014-017-0776-1. PMID 28249612